CLINICAL TRIAL: NCT06463210
Title: Virtual Reality for Pain Management and Patient Satisfaction During Outpatient Hysteroscopy: a Randomized Controlled Trial
Brief Title: Virtual Reality for Pain Management and Patient Satisfaction During Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRHSC 21/278
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Pain, Acute; Satisfaction, Patient
Keywords: Hysteroscopy
MeSH Terms: conditions — Acute Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: 2 randomized groups with 60 patients per arm
Masking Description: Blinding of participants or care providers was not feasible to implement due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse support during hysteroscopy: control group (No Intervention): In our standard hysteroscopy protocol, all patients are advised to take an Ibuprofen 400-600mg or Paracetamol 650-1000 mg two hours before the procedure. They are also suggested to take Bromazepam 1.5 mg two hours before the procedure if they feel anxious.
  As part of our standard procedure during the OH, a trained nurse with >10 years of experience provides distraction and emotional support to the woman. She explains the patient how to breathe and what to expect during the different moments of the procedure, thus involving the women directly in what is happening during the procedure.
- Virtual reality during hysteroscopy: study group (Experimental): In our standard hysteroscopy protocol, all patients are advised to take an Ibuprofen 400-600mg or Paracetamol 650-1000 mg two hours before the procedure. They are also suggested to take Bromazepam 1.5 mg two hours before the procedure if they feel anxious.
  A 360º video was administered to the study group through an Oculus Quest 2™ headset (Meta Platforms, CA. USA). The video was administered through the headset just before the start of the procedure. The video chosen showed a gondola ride through the canals of Venice with relaxing music played on the headset
  Interventions: Device: Virtual reality as a distraction technique

INTERVENTIONS:
Device: Virtual reality as a distraction technique — A 360º relaxing video with music was displayed through a VR headset
  Arms: Virtual reality during hysteroscopy: study group

SUMMARY:
The investigators conducted a randomized controlled trial in 120 patients undergoing an outpatient hysteroscopy (OH).

60 patients were randomly allocated to the control group and 60 patients were randomly allocated to the study group.

The intervention in the study group was to use a virtual reality (VR) device (Meta Quest2) as a distraction technique during the OH.

The investigators wanted to study if the distraction generated by the VR could improve patients' perceived pain or satisfaction with the OH

DETAILED DESCRIPTION:
The investigators conducted a randomized controlled trial in 120 patients undergoing an outpatient hysteroscopy (OH).

60 patients were randomly allocated to the control group and 60 patients were randomly allocated to the study group.

In the standard hysteroscopy protocol, all patients are advised to take an Ibuprofen 400-600mg or Paracetamol 650-1000 mg two hours before the procedure. They are also suggested to take Bromazepam 1.5 mg two hours before the procedure if they feel anxious.

The standard care group had a trained nurse providing distraction and emotional support.

The study group had a VR device (Meta Quest 2) with a video consisting of a gondola ride through the canals of Venice with relaxing music played on the headset The investigators wanted to study if the distraction generated by the VR could improve patients' perceived pain or satisfaction with the OH, comparing it with the standard care group.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive women candidates to undergo an OH
* Women aged 18 to 70 years old

Exclusion Criteria:

* Visual impairment
* Hearing impairment
* Language barrier impeding the correct explanation of the study
* Contraindication for using the VR device
* Confirmed malignant endometrial disease
* Anatomical characteristics impeding the office hysteroscopy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Peak pain | 5-10 minutes after the procedure
  a Visual analogue score (VAS score) between 0 and 10, patients reported their peak perceived pain during the procedure, being 0 no pain and 10 worst pain imaginable
Mean pain | 5-10 minutes after the procedure
  a VAS score between 0 and 10, patients reported their mean perceived pain during the procedure worst pain imaginable

SECONDARY OUTCOMES:
Patient satisfaction with the information received | 5-10 min before the procedure
  Prior to the OH all patients were interrogated about their perception of the information received about the procedure through the question "How has been the information received about the procedure?" (Not enough/Normal/Very good
Patient overall satisfaction with the procedure (OH) | 5-10 min after the procedure
  Overall satisfaction with the OH was assessed through a question formulated as follows: "What is your level of satisfaction with the hysteroscopic procedure?", where patients could evaluate their opinion on a 5-point scale (Very satisfied, Fairly satisfied, Neutral, Somewhat unsatisfied, Very unsatisfied
Patient satisfaction with the VR intervention | 5-10 min after the procedure
  On the study group, patient satisfaction with the VR intervention was also assessed with the following 5-point scale satisfaction question "What is your level of satisfaction with the VR intervention? (Very satisfied, Fairly satisfied, Neutral, Somewhat unsatisfied, Very unsatisfied
Patient satisfaction with the VR intervention | 5-10 min after the procedure
  Patients on the VR group were also asked whether they would like to use the VR if they need to undergo another OH in the future (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
If needed for further studies and with the previous evaluation of the investigators IPD would be available to other researchers

REFERENCES:
- [Background] Vitagliano A, Dellino M, Favilli A, D' Amato A, Nicoli P, Lagana AS, Noventa M, Bochicchio MA, Cicinelli E, Damiani GR. Patients' Use of Virtual Reality Technology for Pain Reduction during Outpatient Hysteroscopy: A Meta-analysis of Randomized Controlled Trials. J Minim Invasive Gynecol. 2023 Nov;30(11):866-876. doi: 10.1016/j.jmig.2023.08.427. Epub 2023 Aug 29. PMID 37648150
- [Background] Deo N, Khan KS, Mak J, Allotey J, Gonzalez Carreras FJ, Fusari G, Benn J. Virtual reality for acute pain in outpatient hysteroscopy: a randomised controlled trial. BJOG. 2021 Jan;128(1):87-95. doi: 10.1111/1471-0528.16377. Epub 2020 Jul 22. PMID 32575151
- [Background] Baradwan S, Alshahrani MS, AlSghan R, Alyafi M, Elsayed RE, Abdel-Hakam FA, Moustafa AA, Hussien AE, Yahia OS, Shama AA, Magdy AA, Abdelhakim AM, Badran H. The effect of virtual reality on pain and anxiety management during outpatient hysteroscopy: a systematic review and meta-analysis of randomized controlled trials. Arch Gynecol Obstet. 2024 Apr;309(4):1267-1280. doi: 10.1007/s00404-023-07319-8. Epub 2024 Jan 2. PMID 38165441
- [Background] Cohen N, Nasra LA, Paz M, Kaufman Y, Lavie O, Zilberlicht A. Pain and anxiety management with virtual reality for office hysteroscopy: systemic review and meta-analysis. Arch Gynecol Obstet. 2024 Apr;309(4):1127-1134. doi: 10.1007/s00404-023-07261-9. Epub 2023 Nov 2. PMID 37917158
- [Background] Pelazas-Hernandez JA, Varillas-Delgado D, Gonzalez-Casado T, Cristobal-Quevedo I, Alonso-Bermejo A, Ronchas-Martinez M, Cristobal-Garcia I. The Effect of Virtual Reality on the Reduction of Pain in Women with an Indication for Outpatient Diagnostic Hysteroscopy: A Randomized Controlled Trial. J Clin Med. 2023 May 24;12(11):3645. doi: 10.3390/jcm12113645. PMID 37297840
- [Background] Sewell T, Fung Y, Al-Kufaishi A, Clifford K, Quinn S. Does virtual reality technology reduce pain and anxiety during outpatient hysteroscopy? A randomised controlled trial. BJOG. 2023 Nov;130(12):1466-1472. doi: 10.1111/1471-0528.17550. Epub 2023 May 23. PMID 37218438
- [Background] Fouks Y, Kern G, Cohen A, Reicher L, Shapira Z, Many A, Yogev Y, Rattan G. A virtual reality system for pain and anxiety management during outpatient hysteroscopy-A randomized control trial. Eur J Pain. 2022 Mar;26(3):600-609. doi: 10.1002/ejp.1882. Epub 2021 Nov 23. PMID 34748679
- [Background] Mirza E, Hanif M, Khan MA, Jaleel S. Re: Virtual reality for acute pain in outpatient hysteroscopy: a randomised controlled trial. BJOG. 2021 Mar;128(4):769-770. doi: 10.1111/1471-0528.16500. Epub 2020 Oct 7. No abstract available. PMID 33027546
- [Derived] Olloqui A, Tejerizo-Garcia A, Guillen C, Perez-Sagaseta C, Gonzalez-Macho C, Bolivar-Miguel AB, Villalba-Gutierrez A, Gil-Ibanez B. Virtual Reality for Pain Management and Patient Satisfaction During Outpatient Hysteroscopy: A Randomised Controlled Trial. BJOG. 2025 Sep;132(10):1416-1425. doi: 10.1111/1471-0528.18228. Epub 2025 May 21. PMID 40400089